CLINICAL TRIAL: NCT01936454
Title: A Study to Evaluate the Contraceptive Effectiveness During the Third, Fourth and Fifth Year of Sino-implant (II) Use and the Pharmacokinetics Over Five Years of Use in Chinese Women
Brief Title: Contraceptive Effectiveness of Sino-implant (II) in China
Status: Completed | Type: Observational
Sponsor: FHI 360 (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 458241-1
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Contraception

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cohort 1: n=20 women with insertion dates 3-5months prior to enrollment and followed for 2-6 months
- Cohort 2: n=20 women with insertion dates 9-11 months prior to enrollment and followed for 2-6 months
- Cohort 3: n=250 women with insertion dates 21-24 months prior to enrollment and followed through month 36
- Cohort 4: n=300 women with insertion dates 33-36 months prior to enrollment and followed through month 6

SUMMARY:
A cohort study to Evaluate the contraceptive effectiveness of Sino-implant (II) during the 3rd and 4th years of use in Chinese women

DETAILED DESCRIPTION:
A Study to Evaluate the Contraceptive Effectiveness during the Third, Fourth and Fifth Year of Sino-implant (II)Use and the Pharmacokinetics (PK) over Five Years of use in Chinese Women

Population: A total of 590 Chinese Sino-Implant (II) users between 20and 44 years of age enrolled in one of four prospective cohorts:

Cohort 1: n=20 women with insertion dates 3-5months prior to enrollment and followed for 2-6 months Cohort 2:n=20 women with insertion dates 9-11 months prior to enrollment and followed for 2-6 months Cohort 3: n=250 women with insertion dates 21-24 months prior to enrollment and followed through month 36 Cohort 4:n=300 women with insertion dates 33-36 months prior to enrollment and followed through month 6

Study Duration: 33 total months in the field: 3 months of participant recruitment(all cohorts); up to 27 months of pregnancy monitoring and PK blood sampling in Cohort 4 (up to 15 months in Cohort 3 and 6 months in Cohort 1 and Cohort 2);and 3 months of close-out activities.

For secondary PK outcomes, blood samples will be taken 2 to 6 months apart from each woman in Cohort 1 and Cohort 2; at enrollment, month 30 and month 36 from the first 20 consenting women in Cohort 3; and at enrollment and months 42, 48, 54, and 60 from the first 30 consenting women in Cohort 4.

Primary Objective: To evaluate the contraceptive effectiveness of Sino-implant (II) during the third and fourth years of use

Secondary Objectives:

1. To evaluate the contraceptive effectiveness of Sino-implant (II) during the fifth year of use.
2. To characterize the total and free levonorgestrel (LNG) plasma concentration-time profiles over five years following Sino-implant (II) insertion
3. To characterize the sex hormone binding globulin (SHBG) serum concentration-time profile and its relationship to total LNG levels over five years following Sino-implant (II) insertion

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed Sino-implant (II) set in place;
* Have a confirmed contraceptive implant insertion date consistent with the criteria for the cohort she is to be enrolled in;
* Be aged between 20 and 44 years, inclusive;
* Not wish to become pregnant in the next year;
* No desire to get implant removal within the next year;
* Be able to understand the information given to them and to make personal decisions on whether to participate or not in the study;
* Consent to participation and sign an informed consent form;
* Agree and be able to return to the clinic for follow-up visit(s).

Exclusion Criteria:

* Acute liver disease or cirrhosis by self-report;
* Benign or malignant tumor of the liver by self-report;
* Use of rifampicin, and/or anticonvulsants (barbiturates, phenytoin, phenobarbital, carbamazepine, oxcarbazepine, primidone, topiramate), and/or herbal products containing St. John's wort (Hypericum perforatum) by self-report;7
* Use of medications containing LNG or other hormones that impact LNG or SHBG disposition, e.g. treatment with LNG or oral contraceptives for bleeding disturbances by self-report;
* Known HIV-positive status by self-report;
* Any condition (social or medical) which in the opinion of the Investigator would make study participation unsafe, would interfere with adherence to study requirements, or complicate data interpretation.

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study Population: Women who have received contraceptive implants from the Tongxiang, An Yang, Lingbao, and Lushi Family Planning Service Stations.
Sampling Method: Non-Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2013-07; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy Pearl Index | 27 months
  Pregnancy Pearl Index (number of pregnancies per 100 woman-years) during the third and fourth years of use, respectively, in Cohort 3 and Cohort 4

SECONDARY OUTCOMES:
Pregnancy Pearl Index during the fifth year of Sino implant (II) use | 27 months
Total and free LNG plasma concentrations measured by a high-performance liquid chromatography with mass spectrometry assay | 27 months
Serum SHBG concentrations measured by a chemiluminescence immunoassay | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Steiner, Ph.D., Principal Investigator — FHI 360
Locations (5):
- China (5):
  - An Yang Population and Family Planning Service Station, Anyang
  - Lingbao Population and Family Planning Service, Lingbao
  - Lushi Family Planning Technical Service Station, Lushi
  - Shanghai Institute of Planned Parenthood, Shanghai
  - Tongxiang Population and Family Planning Service Station, Tongxiang

IPD SHARING:
Plan to Share IPD: Undecided